CLINICAL TRIAL: NCT03982069
Title: Immunological Response to Influenza Vaccination in Children, Adolescents, and Young Adults: A RCT of FluMist vs. Flucelvax
Brief Title: Immunologic Response to FluMist vs. Flucelvax
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Richard Zimmerman MD (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Richard Zimmerman MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY19040242; 1U01|P001035-01 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Influenza, Human; Immune Response
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- FluMist live attenuated influenza vaccine (Active Comparator): Participants receiving live attenuated FluMist influenza vaccine will receive 0.2 mL given intranasally
  Interventions: Biological: FluMist live attenuated influenza vaccine
- Flucelvax inactivated influenza vaccine (Active Comparator): Participants receiving inactivated Flucelvax influenza vaccine will receive 0.5 mL given intramuscularly
  Interventions: Biological: Flucelvax inactivated influenza vaccine

INTERVENTIONS:
Biological: FluMist live attenuated influenza vaccine — Participants randomized to this study influenza vaccine arm will receive FluMist live attenuated influenza vaccine at baseline after the baseline blood draw is complete.
  Arms: FluMist live attenuated influenza vaccine
Biological: Flucelvax inactivated influenza vaccine — Participants randomized to this study influenza vaccine arm will receive Flucelvax cell-culture inactivated influenza vaccine at baseline after the baseline blood draw is complete.
  Arms: Flucelvax inactivated influenza vaccine

SUMMARY:
The purpose of this study is to evaluate immunologic response to different types of influenza vaccine among children/adolescents/young adults 4-21 years of age. This is a randomized controlled trial (RCT), that will assess immune response in about 440 participants (about 220 per vaccine arm) pre- and post-vaccination to FluMist (live attenuated influenza vaccine given by nasal administration) and Flucelvax (egg-free cell-culture inactivated influenza vaccine).

DETAILED DESCRIPTION:
This is a non-blinded, randomized controlled trial analyzing influenza vaccine immunogenicity response in children/adolescents/young adults aged 4-21 years given one of two FDA approved and licensed influenza vaccines: FluMist (live attenuated influenza vaccine by nasal administration) and Flucelvax (egg-free cell-culture inactivated influenza vaccine). This study will enroll about 440 healthy participants, about 220 per vaccine arm. Participants will be randomized in blocks of 4 using a 1:1 allocation to receive either FluMist or Flucelvax. Blood work will be conducted on all participants at baseline prior to vaccine receipt and post-vaccination at Day 7 (range 6-9 days) and Day 28 (range 21-35 days). The primary objective of the study is to determine pre- and post-serologic responses to each vaccine type.

ELIGIBILITY:
Inclusion Criteria:

* aged 4-21 years;
* has prior vaccination history available (which can be determined based either on medical record review or through state registry review);
* plans to receive the current seasonal influenza vaccination at one of the recruiting sites

Exclusion Criteria:

* unable or unwilling to completed required study activities, including informed consent, randomization to vaccine, and bloodwork;
* has already received influenza vaccine for the current season;
* has a known immunocompromising condition or is on an immunosuppressing medication (e.g., high dose steroids >10 days);
* is known to be pregnant;
* has a history of severe allergy to eggs or to influenza vaccine or any of its components

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 465 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Zimmerman, MD, MPH, MA, Principal Investigator — University of Pittsburgh, School of Medicine, Dept. Family Medicine
Locations (2):
- United States (2):
  - General Academic Pediatrics, Pittsburgh, Pennsylvania
  - University of Pittsburgh Department of Family Medicine, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary article, after deidentification, will be placed at the site mentioned below.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months after article publication.
Access Criteria: Researchers who provide a methodologically sound proposal and have appropriate data security and privacy plans in place
URL: http://github.com/pittvax

REFERENCES:
- [Derived] Williams KV, Li ZN, Zhai B, Alcorn JF, Nowalk MP, Levine MZ, Kim SS, Flannery B, Moehling Geffel K, Merranko AJ, Collins M, Susick M, Clarke KS, Zimmerman RK, Martin JM. A Randomized Controlled Trial to Compare Immunogenicity to Cell-Based Versus Live-Attenuated Influenza Vaccines in Children. J Pediatric Infect Dis Soc. 2023 Jun 30;12(6):342-352. doi: 10.1093/jpids/piad033. PMID 37232430

RESULTS

PARTICIPANT FLOW:
Groups:
- FluMist Live Attenuated Influenza Vaccine 2019; FluMist Live Attenuated Influenza Vaccine 2020: Participants receiving live attenuated FluMist influenza vaccine will receive 0.2 mL given intranasally
  FluMist live attenuated influenza vaccine: Participants randomized to this study influenza vaccine arm will receive FluMist live attenuated influenza vaccine at baseline after the baseline blood draw is complete.
- Flucelvax Inactivated Influenza Vaccine 2019; Flucelvax Inactivated Influenza Vaccine 2020: Participants receiving inactivated Flucelvax influenza vaccine will receive 0.5 mL given intramuscularly
  Flucelvax inactivated influenza vaccine: Participants randomized to this study influenza vaccine arm will receive Flucelvax cell-culture inactivated influenza vaccine at baseline after the baseline blood draw is complete.
Period: Overall Study
Arm/Group | FluMist Live Attenuated Influenza Vaccine 2019 | Flucelvax Inactivated Influenza Vaccine 2019 | FluMist Live Attenuated Influenza Vaccine 2020 | Flucelvax Inactivated Influenza Vaccine 2020
Started | 108 | 110 | 127 | 120
Completed | 98 | 100 | 118 | 112
Not Completed | 10 | 10 | 9 | 8
Not completed — Lost to Follow-up | 5 | 5 | 3 | 5
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 5 | 2
Not completed — Specimen loss | 3 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluMist Live Attenuated Influenza Vaccine 2019 | Flucelvax Inactivated Influenza Vaccine 2019 | FluMist Live Attenuated Influenza Vaccine 2020 | Flucelvax Inactivated Influenza Vaccine 2020 | Total
Number analyzed (Participants) | 108 | 110 | 127 | 120 | 465
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47 | 56 | 76 | 74 | 253
  Between 18 and 65 years | 61 | 54 | 51 | 46 | 212
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.8 (4.6) | 16.6 (4.2) | 15.6 (5.0) | 15.1 (5.2) | 16.0 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 71 | 57 | 59 | 254
  Male | 41 | 39 | 70 | 61 | 211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 6 | 4 | 23
  Not Hispanic or Latino | 99 | 104 | 120 | 116 | 439
  Unknown or Not Reported | 2 | 0 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 6 | 7 | 4 | 5 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 43 | 41 | 33 | 21 | 138
  White | 45 | 51 | 79 | 84 | 259
  More than one race | 10 | 9 | 6 | 9 | 34
  Unknown or Not Reported | 4 | 2 | 4 | 1 | 11
Region of Enrollment [Number; unit: participants]
  United States | 108 | 110 | 127 | 120 | 465

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroconversion Response In 2019
Description: Rows in data tables represent different influenza antigens measured in 2019. Hemagglutination inhibition (HI) assay was conducted to assess immunologic outcome. Seroconversion is defined as a 4-fold or higher rise in HI titer post-vaccination given a pre-vaccination HI titer of >=10 and a final HI titer of >=40.
Time Frame: Post-vaccination (at Day 28 timepoint)
Population: 2019 Participants
Measure: Count of Participants; unit: Participants
Arm/Group | FluMist Live Attenuated Influenza Vaccine 2019 | Flucelvax Inactivated Influenza Vaccine 2019
Number analyzed (Participants) | 98 | 100
Participants
  A/H1N1-A/Brisbane | 5 | 33
  A/H3N2-A/Kansas egg grown virus | 11 | 44
  A/H3N2-A/Kansas cell grown virus | 8 | 47
  B/Victoria-B/Colorado | 9 | 28
  B/Yamagata-B/Phuket | 4 | 29
Statistical Analysis 1: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p < 0.001, Chi-squared — All listed antigens

2. Primary Outcome: Number of Participants With Seroconversion Response In 2020
Description: Rows in data tables represent different influenza antigens measured in 2020. Hemagglutination inhibition (HI) assay was conducted to assess immunologic outcome. Seroconversion is defined as a 4-fold or higher rise in HI titer post-vaccination given a pre-vaccination HI titer of >=10 and a final HI titer of >=40.
Time Frame: Post-vaccination (at Day 28 timepoint)
Population: 2020 Participants
Measure: Count of Participants; unit: Participants
Arm/Group | FluMist Live Attenuated Influenza Vaccine 2020 | Flucelvax Inactivated Influenza Vaccine 2020
Number analyzed (Participants) | 118 | 112
Participants
  A/H1N1-A/Hawaii66 egg based antigen | 8 | 59
  A/H1N1-A/Hawaii70 cell based antigen | 10 | 58
  A/H1N1-A/Delaware | 2 | 38
  A/H3N2-A/Hong Kong | 14 | 48
  B/Victoria-B/Washington | 13 | 36
  B/Yamagata-B/Phuket | 11 | 32
Statistical Analysis 1: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p < 0.001, Chi-squared — All listed antigens

3. Secondary Outcome: Number of Participants With Seroprotection Response in 2019
Description: Rows in data tables represent different influenza antigens measured in 2019. Hemagglutination inhibition (HI) assay was conducted to assess immunologic outcome. Seroprotection is defined as a HI titer >= 1:110 at either time point.
Time Frame: Pre-vaccination (at Day 0 timepoint) and post-vaccination (at Day 28 timepoint)
Population: 2019 Participants
Measure: Count of Participants; unit: Participants
Arm/Group | FluMist Live Attenuated Influenza Vaccine 2019 | Flucelvax Inactivated Influenza Vaccine 2019
Number analyzed (Participants) | 98 | 100
Participants
  A/H1N1-A/Birsbane:Day 0 | 54 | 61
  A/H1N1-A/Birsbane:Day 28 | 58 | 93
  A/H3N2-AKansas egg grown virus: Day 0 | 34 | 41
  A/H3N2-AKansas egg grown virus: Day 28 | 41 | 77
  A/H3N2-AKansas cell grown virus: Day 0 | 14 | 24
  A/H3N2-AKansas cell grown virus: Day 28 | 26 | 65
  B/Victoria-B/Colorado: Day 0 | 34 | 34
  B/Victoria-B/Colorado: Day 28 | 36 | 71
  B/Yamagata-B/Phuket: Day 0 | 57 | 51
  B/Yamagata-B/Phuket: Day 28 | 57 | 84
Statistical Analysis 1: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p < 0.001, Chi-squared — Day 28 for all listed antigens
Statistical Analysis 2: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p = 0.40, Chi-squared — Day 0, A/H1N1-A/Brisbane
Statistical Analysis 3: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p = 0.36, Chi-squared — Day 0 A/H1N1-A/Kansas egg grown virus
Statistical Analysis 4: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p = 0.08, Chi-squared — Day 0 A/H1N1-A/Kansas cell grown virus
Statistical Analysis 5: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p = 0.91, Chi-squared — Day 0 B/Victoria-B/Colorado
Statistical Analysis 6: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p = 0.31, Chi-squared — Day 0 B/Yamagata-B/Phuket

4. Secondary Outcome: Geometric Mean Titers (GMTs) at Each Time Point 2019
Description: Rows in data tables represent different influenza antigens measured in 2019. Hemagglutination inhibition assay was conducted to assess immunologic outcome. GMTs is defined as the anti-log of the mean of the log2 HI titers
Time Frame: Pre-vaccination (at Day 0 timepoint) and post-vaccination (at Day 28 timepoint)
Population: 2019 Participants
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | FluMist Live Attenuated Influenza Vaccine 2019 | Flucelvax Inactivated Influenza Vaccine 2019
Number analyzed (Participants) | 98 | 100
titer
  A/H1N1-A/Brisbane: Day 0 | 94 [77 to 116] | 90 [73 to 111]
  A/H1N1-A/Brisbane: Day 28 | 108 [89 to 132] | 269 [228 to 317]
  A/H3N2-A/Kansas egg grown virus: Day 0 | 75 [64 to 89] | 78 [66 to 95]
  A/H3N2-A/Kansas egg grown virus: Day 28 | 96 [83 to 112] | 205 [178 to 237]
  A/H3N2-A/Kansas cell grown virus: Day 0 | 50 [43 to 58] | 46 [38 to 55]
  A/H3N2-A/Kansas cell grown virus: Day 28 | 63 [58 to 74] | 136 [113 to 165]
  B/Victoria-B/Colorado: Day 0 | 65 [53 to 81] | 65 [53 to 79]
  B/Victoria-B/Colorado: Day 28 | 78 [64 to 94] | 158 [134 to 186]
  B/Yamagata-B/Phuket: Day 0 | 101 [83 to 122] | 89 [74 to 107]
  B/Yamagata-B/Phuket: Day 28 | 107 [90 to 128] | 215 [191 to 241]
Statistical Analysis 1: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p = 0.79, t-test, 2 sided — Day 0 A/H1N1-A/Brisbane
Statistical Analysis 2: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p = 0.79, t-test, 2 sided — Day 0 A/H3N2-A/Kansas egg grown virus
Statistical Analysis 3: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p = 0.56, t-test, 2 sided — Day 0 A/H3N2-A/Kansas cell grown virus
Statistical Analysis 4: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p = 0.95, t-test, 2 sided — Day 0 B/Victoria-B/Colorado
Statistical Analysis 5: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p = 0.44, t-test, 2 sided — Day 0 B/Yamagata-B/Phuket
Statistical Analysis 6: Comparison: FluMist Live Attenuated Influenza Vaccine 2019 vs Flucelvax Inactivated Influenza Vaccine 2019; Test type: Other; p < 0.001, t-test, 2 sided — Day 28 for all listed variables

5. Secondary Outcome: Number of Participants With Seroprotection Response in 2020
Description: Rows in data tables represent different influenza antigens measured in 2020. Hemagglutination inhibition (HI) assay was conducted to assess immunologic outcome. Seroprotection is defined as a HI titer >= 1:110 at either time point.
Time Frame: Pre-vaccination (at Day 0 timepoint) and post-vaccination (at Day 28 timepoint)
Population: 2020 Participants
Measure: Count of Participants; unit: Participants
Arm/Group | FluMist Live Attenuated Influenza Vaccine 2020 | Flucelvax Inactivated Influenza Vaccine 2020
Number analyzed (Participants) | 118 | 112
Participants
  A/H1N1-A/Hawaii66 egg: Day 0 | 25 | 25
  A/H1N1-A/Hawaii66 egg: Day 28 | 33 | 79
  A/H1N1-A/Hawaii70 cell grown virus: Day 0 | 59 | 54
  A/H1N1-A/Hawaii70 cell grown virus: Day 28 | 65 | 102
  A/H1N1-A/Delaware: Day 0 | 37 | 32
  A/H1N1-A/Delaware: Day 28 | 43 | 65
  A/H3N2-A/Hong Kong: Day 0 | 90 | 73
  A/H3N2-A/Hong Kong: Day 28 | 102 | 99
  B/Victoria-B/Washington: Day 0 | 62 | 59
  B/Victoria-B/Washington: Day 28 | 71 | 86
  B/Yamagata-B/Phuket: Day 0 | 66 | 54
  B/Yamagata-B/Phuket: Day 28 | 64 | 92
Statistical Analysis 1: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.83, Chi-squared; Day 0: A/H1N1-A/Hawaii66-egg based antigen
Statistical Analysis 2: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.79, Chi-squared; Day 0: A/H1N1-A/Hawaii70-cell based antigen
Statistical Analysis 3: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.65, Chi-squared; Day 0: A/H1N1-A/Delaware
Statistical Analysis 4: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.06, Chi-squared; Day 0: A/H3N2-A/Hong Kong
Statistical Analysis 5: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.98, Chi-squared; Day 0: B/Victoria-B/Washington
Statistical Analysis 6: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.24, Chi-squared; Day 0: B/Yamagata-B/Phuket
Statistical Analysis 7: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p < 0.01, Chi-squared; Day 28: A/H1N1-A/Hawaii66-egg based antigen, A/H1N1-A/Hawaii70-cell based antigen, A/H1N1-A/Delaware, B/Victoria-B/Washington, B/Yamagata-B/Phuket
Statistical Analysis 8: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.66, Chi-squared; A/H3N2-A/Hong Kong

6. Secondary Outcome: Geometric Mean Titers (GMTs) at Each Time Point 2020
Description: Rows in data tables represent different influenza antigens measured in 2020. Hemagglutination inhibition assay will be conducted to assess immunologic outcome. GMTs is defined as the anti-log of the mean of the log2 HI titers
Time Frame: Pre-vaccination (at Day 0 timepoint) and post-vaccination (at Day 28 timepoint)
Population: 2020 Participants
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | FluMist Live Attenuated Influenza Vaccine 2020 | Flucelvax Inactivated Influenza Vaccine 2020
Number analyzed (Participants) | 118 | 112
titer
  A/H1N1-A/Hawaii66 egg grown virus: Day 0 | 42 [33 to 52] | 34 [27 to 43]
  A/H1N1-A/Hawaii66 egg grown virus: Day 28 | 51 [41 to 63] | 171 [139 to 211]
  A/H1N1-A/Hawaii70 cell grown virus: Day 0 | 97 [80 to 118] | 84 [61 to 103]
  A/H1N1-A/Hawaii70 cell grown virus: Day 28 | 121 [100 to 145] | 380 [315 to 458]
  A/H1N1-A/Delaware: Day 0 | 58 [47 to 72] | 46 [36 to 57]
  A/H1N1-A/Delaware: Day 28 | 62 [50 to 78] | 120 [100 to 145]
  A/H3N2-A/Hong Kong: Day 0 | 174 [133 to 226] | 119 [89 to 160]
  A/H3N2-A/Hong Kong: Day 28 | 234 [190 to 288] | 370 [282 to 484]
  B/Victoria-B/Washington: Day 0 | 92 [75 to 114] | 88 [70 to 111]
  B/Victoria-B/Washington: Day 28 | 116 [95 to 142] | 212 [175 to 258]
  B/Yamagata-B/Phuket: Day 0 | 98 [83 to 118] | 87 [71 to 107]
  B/Yamagata-B/Phuket: Day 28 | 114 [96 to 135] | 214 [184 to 249]
Statistical Analysis 1: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.22, t-test, 2 sided — Day 0: A/H1N1-A/Hawaii66 egg based antigen
Statistical Analysis 2: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.25, t-test, 2 sided — Day 0: A/H1N1-A/Hawaii70 cell based antigen
Statistical Analysis 3: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.13, t-test, 2 sided — Day 0: A/H1N1-A/Delaware
Statistical Analysis 4: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.06, t-test, 2 sided — Day 0: A/H3N2-A/Hong Kong
Statistical Analysis 5: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.78, t-test, 2 sided — Day 0: B/Victoria-B/Washington
Statistical Analysis 6: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.36, t-test, 2 sided — Day 0: B/Yamagata-B/Phuket
Statistical Analysis 7: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p < 0.0001, t-test, 2 sided — Day 28: A/H1N1-A/Hawaii66 egg based antigen, A/H1N1-A/Hawaii70 cell based antigen, A/H1N1-A/Delaware, B/Victoria-B/Washington, B/Yamagata-B/Phuket
Statistical Analysis 8: Comparison: FluMist Live Attenuated Influenza Vaccine 2020 vs Flucelvax Inactivated Influenza Vaccine 2020; Test type: Other; p = 0.01, t-test, 2 sided — Day 28: A/H3N2-A/Hong Kong

ADVERSE EVENTS:
Time Frame: 5 weeks in relation to baseline
Arm/Group | FluMist Live Attenuated Influenza Vaccine | Flucelvax Inactivated Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 0/235 | 0/230
Serious Adverse Events (participants affected / at risk) | 0/235 | 0/230
Other Adverse Events (participants affected / at risk) | 0/235 | 0/230

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT03982069/Prot_SAP_ICF_000.pdf